CLINICAL TRIAL: NCT05829577
Title: The Effectiveness of Using Daily Living Skills and Sensory Integration Training Combined With Executive Function Strategies for Improving Self-Care, Sensory Integration and Fine Motor Skills in Children With ASD in Qatar: A Randomized Control Trial
Brief Title: Integrated Life Skill Training and Executive Function Strategies in Children With ASD
Acronym: ASD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hamad General Hospital (Other Government)
Collaborators: Universiti Sultan Zainal Abidin (Other)
Responsible Party: Principal Investigator, Bara Yousef, Occupational Therapy Specialist, Hamad General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MRC-01-22-509
Record Dates: First submitted 2023-04-01; First posted 2023-04-25 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Autism Spectrum Disorder
Keywords: ASD
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: Single blind one center randomized control trial (RCT) with one arm :control group will receive Individual Sensory integration / sensory processing and daily life skills training , treatment group will receive Individual Sensory integration / sensory processing and daily life skills training training combined with EF strategies both groups will receive 1 session individual OT/week for 45 min for 14 weeks .
Who Masked: Outcomes Assessor
Masking Description: Administration of assessment will be done by(individuals blinded of the outcome assessor) as an Independent evaluators, whose trained in the administration of study assessments, will conduct the pre-intervention, re assessment and post intervention assessments and this therapist will be blinded for intervention and control group, and thire qualification as follow : highly experienced therapist who has been licensed to practice occupational therapy for a mean of 10 years, and who had experience with working with children with ASD (mean = 5 years). also were trained on conducting these standardized assessment and certified on Wee FIM
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Executive function treatment (Experimental): Patient will receive Individual DLS and SI/SP training combined with EF strategies
  Interventions: Other: Executive Function Strategies and Training; Other: Daily Life skill training; Other: Sensory Integration /Processing training
- Treatment as usual (Active Comparator): patient will receive Individual DLS and SI/SP training.
  Interventions: Other: Daily Life skill training; Other: Sensory Integration /Processing training

INTERVENTIONS:
Other: Executive Function Strategies and Training — will be conducted by primary investigator and trained therapist ,EF strategies will be implemented during DLS and SI training and these strategies will target following area which proved by evidences within the context of functional training: Using monitoring system for each child , Improving sense of time, Externalize important information , Externalize Motivation, Provide consequences: Immediately, more frequently, Higher magnitude and more powerful, Richer degree of incentive, Rotated or changed more frequently, Personalize the command, praise, instruction, reprimanding, Process training, remediation and training on executive function skill
  Arms: Executive function treatment
Other: Daily Life skill training — each child will receive 25 minute of DLS training which will focus on training children on Grooming, feeding, dressing undressing, toileting and community reintegration tasks aligned with facilitation fine motor skills for children and Using several techniques for ADL training including : prompting, shaping, forward and backward chaining, and modeling ,training children based on level of independency identified by WeeFIM score
Other: Sensory Integration /Processing training — each patient will receive 20 min of SI/SP training Manualized SI/SP intervention which will be used is based on the principles of sensory integration as outlined by Ayres ,such as deep pressure, brushing, weighted vests, and swinging will used , individually-tailored treatment activities might include activities such as using a carpeted scooter board while in the prone position to pull oneself up a ramp, then working to turn the scooter board around to ride down the ramp and land in a cushioned area of mats and pillows that are covered with various textures. Intervention is contextualized in play with active involvement of the child will be conducted in a large gym equipped with mats, a variety of suspended swings, large balls, a climbing wall, carpeted barrels, large inner tubes and foam blocks with opportunities for active, guided, sensory motor play.

SUMMARY:
The goal of this clinical trial is to test if using what is called executive function strategies like strategies for improving self-regulation ,strategies for improving planning and problem solving work well when applied within occupational therapy treatment program for children who is diagnosed with Autism Spectrum Disorder , the study will compare between applying regular occupational therapy alone and applying regular occupational therapy plus executive function strategies in improving children with autism spectrum disorder , they will be two group in the study: first group called control group and second group called intervention group, if child is assign on control group he/she will receive regular individual occupational therapy services in autism program which is :Sensory integration which might include things like playing with different interactive games, different textures swinging, bouncing or climbing , and children will also receive life skill training which target training child on self-care skill like grooming, feeding, dressing undressing and toiling skills ) And (if the child assigned on intervention group he/she will receive also regular individual occupational therapy services which described above plus getting executive function training which will be implemented during training the child on daily life skill and this might include using timer during the training, organized schedules, special motivation system and others ,before enrolling children on treatment or control group parent will be asked to sign consent form and after that children will screened based on specific criteria make sure that they are fit for the study then if they meet the study criteria they will also "randomized" into one of two study groups ,Randomization means that putting child into a group by chance. It is like flipping a coin and each child will have a 50% chance of being place in a specific group, following that children will be have detailed assessments which will be done by an experienced occupational therapist and these assessment is aiming to measure the improvement on children condition after receiving therapy ,and will done before treatment , after seven weeks of treatment and completion program at 14 week then data from assessment will be analyzed, each group will receive forty five min regular weekly individual therapy sessions and this extent for thirteen weeks .

DETAILED DESCRIPTION:
The goal of this clinical trial is to test if using what is called executive function strategies like strategies for improving self-regulation ,strategies for improving planning and problem solving work well when applied within occupational therapy treatment program for children who is diagnosed with Autism Spectrum Disorder , the study will compare between applying regular occupational therapy alone and applying regular occupational therapy plus executive function strategies in improving children with autism spectrum disorder , regular occupational therapy consist of 1. Sensory integration and sensory processing Training which target reduction of sensory problem those children might like : sensitivity to sound or lights, selective and picky eating, hypersensitivity to touch and different texture, avoidant of some body movement or hyperactivity, 2.Dailiy life skills Training : like training children on grooming skills, dressing and undressing and toilet training ,and the main question which aim to answer : Is the use of Executive strategies combined with training Sensory integration / sensory processing and daily life skills training more effective than Sensory integration and daily life skill training alone in improving children with Autism Spectrum Disorder ? they will be 2 group in the study: first group called control group and second group called intervention group, if child is assign on control group he/she will receive regular individual occupational therapy services in autism program which is :Sensory integration therapy which involve activities to stimulate sensory responses from the child ,this might include things like playing with different interactive games, different textures swinging, bouncing or climbing , and child will also receive life skill training which target training child on self-care skill like grooming, feeding, dressing undressing and toiling skills ) And (if the child assigned on intervention group he/she will receive also regular individual occupational therapy services which described above plus getting executive function training which will be implemented during training the child on daily life skill and this might include using timer during the training, organized schedules, special motivation system and others which will be explained in more details by therapist before commencing with treatment .

before enrolling children on treatment or control group parent will be asked to sign consent form and after that children will screened based on specific criteria make sure that they are fit for the study then if they meet the study criteria they will also "randomized" into one of two study groups ,Randomization means that you are put into a group by chance. It is like flipping a coin and each child will have a 50% chance of being place in a specific group, following that children will be have detailed assessments which will be done by an experienced occupational therapist and these assessment is aiming to measure the improvement on child condition after receiving therapy ,and will done before treatment and after seven weeks of treatment and after completion of treatment and after completion all dat from these assessments will analyzed , each group will receive forty five min regular weekly individual therapy sessions and this extent for thirteen weeks .

Primacy outcome measure will be :

1. Verbal Behavior Milestones Assessment and Placement Program (VB-MAPP) will be used for determining the inclusion criteria and measuring improvement on self help skills,
2. Pediatric Functional Independent Measure (WeeFIM): will be used to measure improvement in self-care and social cognition skills,
3. Short Sensory Profile™ 2 (SSP2) will be used to measure improvement in sensory processing , Sp2 comprise 34-item caregiver questionnaire

Secondary Outcome measure will be :

Visual Motor Integration Test (Beery-VMI) will be used to monitor changes in visual motor integration skills as part of fine motor skills Primary outcome of the study will be measured based on (VB-MAPP,SP2,VMI,WeeFIM) Changes in the pretest-and posttest scores(Standard Score, Percentile Rank, P value) will be compared between the intervention and control groups using a Linear-mixed regression model and analysis of covariance (ANCOVA)Using repeated-measures analysis of variance, with comparing baseline scores with reassessment and poste treatment scores.

To analyze the data, Statistical Package for Social Science (SPSS-28) software will be used.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were diagnosed with ASD
* Those who were referred to Autism Program
* Those aged 3-5 years (Diamond, 2013)
* Patients first admitted to Autism Individual therapy program .
* All children with different language will be included and if parents couldn't complete some of the required outcome measure, they will be excluded on the analysis stage of study

Exclusion Criteria:

* Patients who have severe Impairment learning and linguistic acquisition skill based on VB-MAPP (has score 4 on any item of Barrier Assessment)
* Those who did not provide consent for the study

Elimination criteria

* Children who do not complete 13 intervention sessions following the research protocol .
* Children who received other interventions that may affect the study results .

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 92 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-08-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Verbal Behavior Milestones Assessment and Placement Program (VB-MAPP) | Will be done before treatment ,after 7 week of treatment , and after treatment completion at 14 week
  will be used for determining if participant is eligible for study and measuring change on self help skills.
Pediatric Functional Independent Measure (WeeFIM) | Will be done before treatment ,after 7 week of treatment , and after treatment completion at 14 week
  will be used to measure changes in self-care and social cognition skills .
Short Sensory Profile™ 2 (SSP2) | Will be done before treatment ,after 7 week of treatment , and after treatment completion at 14 week
  will be used to measure improvement in sensory processing skills .

SECONDARY OUTCOMES:
Visual Motor Integration Test (Beery-VMI) | Will be done before treatment ,after 7 week of treatment , and after treatment completion at 14 week
  will be used to monitor changes in visual motor integration skills as part of fine motor skills

CONTACTS AND LOCATIONS:
Overall Officials: BARA M YOUSEF, Bsc, Principal Investigator — Hamad Medical Corporation
Locations (1):
- Hamad Medical Corporation, Doha, Qatar -doha, Qatar

IPD SHARING:
Plan to Share IPD: No